CLINICAL TRIAL: NCT03495414
Title: Neurobiologisk Bakgrund Till Hypersexuell Störning
Brief Title: Neurobiological Underpinnings to Hypersexual Disorder
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital, ANOVA, Stockholm (Stefan Arver, Katarina Görts Öberg) (Unknown)
Responsible Party: Principal Investigator, Christoph Abé, Assistant Professor, Karolinska Institutet
Other Study IDs: 2017/2152-31
Record Dates: First submitted 2018-03-20; First posted 2018-04-12 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Hypersexuality; Hypersexual Disorder; Compulsive Sexual Behavior
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder | interventions — Neuroimaging; Neuropsychological Tests; Psychometrics; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA extraction is planned for potential epigenetic profiling for analysis of genes related to regulation of the HPA-axis and other relevant epigenomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls (HC): Controls will be physically and psychologically healthy and will show no indication of clinical hypersexuality.
  Interventions: Other: Brain Imaging; Other: Cognitive testing; Other: Psychometric; Other: Blood test
- Patients with hypersexual disorder (HD): Patients will meet diagnostic criteria for HD as defined in the DSM-5 proposed criteria for hypersexual disorder (Kafka, 2010) and CSBD according to ICD-11.
  Interventions: Other: Brain Imaging; Other: Cognitive testing; Other: Psychometric; Other: Blood test

INTERVENTIONS:
Other: Brain Imaging — * Structural MRI (T1 weighted)
  * Diffusion Tensor Imaging (DTI)
  * resting state functional MRI (rs-fMRI)
  * functional MRI (fMRI): Brain activity will be measured in response to sexual images (visually evoked sexual arousal; processing of sexual stimuli), and importantly during a phase when these stimuli are anticipated (neural correlates of wanting and desire; reward anticipation).
Other: Cognitive testing — We will administer neuropsychological tests assessing objective measures for
  * intelligence (Ravens Matrices)
  * impulsivity and risk-taking behavior (Balloon Analogue Risk Task)
  * inhibitory control (Stop Signal Task).
Other: Psychometric — Administered questionnaires include anxiety and depression symptoms (MADRS, HADS, GAD), drug use (AUDIT, DUDIT), attention deficits (ASRS), impulsivity (BIS-11), reward seeking behavior (BIS/BAS), sexual orientation, (hyper)sexual behavior, desire and compulsivity aspects (HDSI, HBI, SCS, SDI, SIS/SES).
Other: Blood test — Blood samples will be taken for routine health assessment, measurement of sex hormonal levels, HPA-axis function test (dexamethasone suppression), and potential DNA extraction and (epi)genetic profiling.

SUMMARY:
Hypersexual Disorder (HD), sometimes called "sexual addiction", is a disorder with intense sexual desires and psychological preoccupations that lead to out-of-control sexual activities with severe consequences. HD is related to higher risks of HIV infection and an important risk factor for committing sexual crimes. The prevalence of HD is 3-6% of the general population, thus, a significant burden for society. The neurobiological mechanisms behind HD are still unknown, and there is still a great need for causal treatments.

This study is aimed at identifying neurobiological and psychological mechanisms underlying HD as a basis for treatment development. The overall goal is to improve mental health, quality of life, diagnosis and treatment options for affected individuals, and to reduce the impact HD can have on society. Patients with HD will be recruited at Karolinska University Hospital in close collaboration between endocrinologists, psychologists, psychiatrists, and brain researchers at Karolinska Institutet. Cases and healthy controls will undergo brain scans (MRI), psychological and blood tests to quantify neurobiological, cognitive, and behavioral aspects of HD.

This study is directly integrated into clinical practice, can identify important targets for interventions and factors predicting treatment outcomes. This study is essential for a better understanding of HD, the improvement of treatments, and can have significant impact on the prevention of HIV infections and sexual crimes.

ELIGIBILITY:
Inclusion Criteria:

* Male
* At least 18 years of age,
* Fluent in the Swedish language
* Patients will meet diagnostic criteria for hypersexual disorder and will not have started with any psychotherapy or psychological treatment.
* Controls will be physically and psychologically healthy, and show no indication of clinical hypersexuality

Exclusion Criteria:

For both patients and controls any reported medical or clinical condition known to affect brain structure and function, test performance, or associated with risks for the MRI environment will be exclusionary. The investigators will exclude for the following:

* Severe neurological/psychiatric diseases or conditions (e.g., major depression, bipolar disorder, ADHD, autism, anxiety/panic disorder, obsessive compulsive disorder, personality disorder, Parkinson's disease, epilepsy, PTSD/chronic stress/burnout syndrom, Alzheimer's disease)
* Gender identity disorder/gender dysphoria
* Chronic pain conditions
* Impared vision, or other vision problems that cannot be corrected with MR-safe equipment.
* Hearing impairments, or problems with other senses
* History of severe brain damage/injuries
* Claustrophobia
* Having metal implants, a pacemaker, metallic braces or other MRI contra-indications
* Alcohol/drug dependence/abuse, eating disorder, pathological gambling, during the past 6 months.
* HIV and Hepatitis C/B, if the condition is untreated or virus levels detectable.
* Untreated endocrinologic diseases
* Medication: bensodiazepine, antipsychotics, mood stabilizers, centrally acting sympathicomimetics, SSRI (if use started less than 3 months ago). Any medication or pharmaceutical drug that interferes with sex hormone production or metabolism, i.e. ketoconazol, cyproteronacetate, spironolactone and similar drugs.

Note: There is a potentially higher prevalence of comorbidities and medication use in patients. To facilitate recruitment and study completion, the investigators may include subjects that report specific conditions at the discretion of the principle investigator. In those cases, corresponding information will be recorded in order to control for potential confounders.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to known effects on brain structure and function, gender dysphoria is an exclusionary condition in this part of the study.
Study Population: Patients will be recruited through an ongoing CBT study (KAFKA_IT) at Karolinska University Hospital (ANOVA). Initial contact between patients and study coordinators will primarily be made through the phone helpline PrevenTell, designed to prevent sexual offences by targeting persons at risk. At the clinical visit patients will be evaluated in a face to face interview by trained psychologists/psychiatrists to establish psychiatric diagnoses, including the diagnosis of HD. If criteria for HD are met, patients will be informed about the present imaging study. Healthy controls from the Stockholm catchment area will be recruited through Karolinska Trial Alliance, and/or public advertisement in form of posters, online job postings and/or social media.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Brain activity | acquired during brain imaging experiment (MRI scan day)
  Functional brain response (BOLD activity) upon presentation and anticipation of visual sexual stimuli.
Anatomical brain measures | Acquired during brain imaging experiment (MRI scan day)
  Measures for brain morphology (regional cortical volume, thickness, surface area, and subcortical volumes)

SECONDARY OUTCOMES:
Resting state fMRI | Acquired during fMRI experiment (MRI scan day)
  Functional connectivity
Diffusion MRI | Acquired during fMRI experiment (MRI scan day)
  Structural connectivity
Reaction times | Acquired during fMRI experiment (MRI scan day)
  Response reaction times during fMRI task
Raven Progressive Matrices (cognitive task) | Acquired at brain MRI assessment day, or as close to this day as possible.
  Objective measures for intelligence
Balloon Analogue Risk Task (cognitive task) | Acquired at brain MRI assessment day, or as close to this day as possible.
  Objective measures for impulsivity/risk-taking
Stop Signal Task (cognitive task) | Acquired at brain MRI assessment day, or as close to this day as possible.
  Objective measures for inhibitory control
MADRS-S (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Montgomery Asberg Depression Rating Scale
ASRS (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Adult ADHD Self-Report Scale
AUDIT (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Alcohol Use Disorders Identification Test
DUDIT (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Drug Use Disorders Identification Test
EQ-5D (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  General Health information
4-item Kinsey-scale (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Sexual Orientation Dimension
HDSI (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Hypersexual Disorder Screening Inventory
SCS (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Sexual Compulsivity Scale
HBI (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Hypersexual Behavior Inventory
SIS/SES (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Sexual Inhibition/Excitation Scale
HADS (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Hospital Anxiety and Depression Scale
GAD (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  General Anxiety Disorder scale
BRSI-SE (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Bem Sex Role Inventory
RAADS (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Ritvo Autism Asperger Diagnostic Scale
SDI (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Sexual Desire Inventory
BIS-11 (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Barratt Impulsiveness Scale
BIS/BAS (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Behavioral Inhibition/Activation System
Sexual Behavior (questionnaire) | Assessed through an online platform (as close to MRI scan day), and/or at MRI scan day
  Frequency of pornography consumption and sexual encounters.
fMRI experience rating (questionnaire) | Assessed right before and after MRI scan
  Ratings of emotions experienced in context of the fMRI task, incl. craving/desire, stimuli induced sexual arousal.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital (ANOVA), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided